CLINICAL TRIAL: NCT05291793
Title: The Effect of Different Intra-articular Injections on Pain and Function in Primary Gonarthrosis
Brief Title: The Effect of Different Intra-articular Injections Primary Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Yiğit Umur Cırdı, Medical Doctor, Orthopedics and Traumatolgy Specialist, Principal Investigator, Acibadem Kozyatagi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2100027722
Record Dates: First submitted 2022-02-25; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Gonarthrosis; Primary
Keywords: Gonarthrosis; Saline injection; intra-articular
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — tenoxicam; Powders; Solutions; Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Identical work scheme applied in 4 different centers by 4 Physicians. Both patient selection, randomization, and blind injection applications have been implemented in same order.
Who Masked: Participant, Care Provider
Masking Description: patients were not aware of the ingredient of the injection they had received Care providers were not aware of the ingredient of injection during application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NSAID group (No Intervention): Group 1, patients only received non-steroid anti-inflammatory oral and topical treatment for 3 weeks. (ibuprofen 2x800 mg (1600 mg daily), 1% nimesulide + 5%Lidocain (3 times a day))
- Tenoxicam (Active Comparator): Group 2, patients received intraarticular tenoxicam ( 20 mg) once.
  Interventions: Drug: Tenoxicam 20 Mg Powder for Solution for Injection Vial
- Methylprednisolone (Active Comparator): Group 3, patients received intraarticular methylprednisolone once(40mg).
  Interventions: Drug: Methylprednisolone
- Saline (Sham Comparator): Group 4, patients received an intraarticular sterile saline injection(4ml).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tenoxicam 20 Mg Powder for Solution for Injection Vial — Tenoxicam 20 Mg Powder is mixed with dissolving solvent then administered intraarticularly
  Arms: Tenoxicam
Drug: Methylprednisolone — Methylprednisolone 40 Mg (suspension) administered intraarticularly
  Arms: Methylprednisolone
Drug: Saline — 2ml sterile saline administered intraarticularly
  Arms: Saline

SUMMARY:
Gonarthrosis is a frequent cause of knee pain and mostly related to altered function of the knee. Intra-articular injections are a valuable noninvasive medical treatment of choice for pain management and functional enhancement. This study aims to investigate the effects of intra-articular injections without local anesthesics which are well known to be chondrotoxic. For this purpose, functional data of the patients who received intra-articular injections have been collected and analyzed.

DETAILED DESCRIPTION:
Intra-articular knee injections are commonly used treatment method. It is preferred to relieve the pain and functional limitation due to knee osteoarthritis. Studies have shown the benefit of intra-articular injections, including intra-articular sterile saline injection alone. In addition, studies have shown chondrotoxic effects of local anesthetics and corticosteroids such as triamcinolone. Local anesthetics are often added to the injection in intra-knee injections. Many previous studies stated that anesthetic agents were mixed with corticosteroid and NSAID intra-articular injections but not in this study. This creates confusion on which preparation is effective on pain and function. The aim of this study is to compare pain-reducing and function-improving effects of intra-articular injection with corticosteroids or NSAIDs, while avoiding local anesthetics whose chondrotoxic effects have been confirmed. In order to reveal the unmasked effect, an intra-articular saline injection group was introduced as a sham treatment. Thus, a study with a level of evidence 1 will make a significant contribution to the literature.

Patients who applied to the outpatient clinic and who were diagnosed with primary gonarthrosis by clinical and radiographic examinations have been randomized to four different groups by closed-envelope method following taking the informed consent. Accordingly, nonsteroidal anti-inflammatory (NSAI) drugs have been prescribed to all diagnosed patients. Demographic data of the patients have been noted and randomized into four equal groups of thirty individuals each. Afterwards, the first group received NSAID treatment, the second group received intra-articular methylprednisolone, the third group received intraarticular tenoxicam, and the fourth group received intra-articular sterile saline injection. All eligible patients have been given one random envelope by the secretary, then proceeded to the injection room with envelopes closed. The orthopedic technician prepared the injection depending on the information inside the envelope then the syringe is covered with opaque plaster or foil. Then, an injection was applied by the physician blindly. The patients' visual analog score(VAS) pain form and WOMAC scores are collected in each follow-up. Following the data has been obtained by an independent data recorder, all data have been saved to the database and statistical results were analyzed. According to the posthoc power analysis, the number of patients can be revised for statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Diagnosed as Osteoarthritis ( in weight-bearing standing Antero-Posterior and Lateral knee plain radiographs)

Exclusion Criteria:

* Patients refuse to enroll in the study voluntarily
* Patients refuse to give informed consent
* Patients who have received physiotherapy and/or intraarticular injection in the last 6 months.
* Patients who have used supporting brace treatment in the last 6 months
* Patients did not attend routine follow-up visits.
* Patients experienced any allergic reaction to the administered drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks prior to intra-articular injection
  Visual Analogue Scale ( Score:0 corresponds to 'no pain', score:10 corresponds to excessive pain)
Visual Analogue Scale (VAS) | at 2nd week following intra-articular injection
  Visual Analogue Scale ( Score:0 corresponds to 'no pain', score:10 corresponds to excessive pain)
Visual Analogue Scale (VAS) | at 4th week following intra-articular injection
  Visual Analogue Scale ( Score:0 corresponds to 'no pain', score:10 corresponds to excessive pain)
Visual Analogue Scale (VAS) | at 6th week following intra-articular injection
  Visual Analogue Scale ( Score:0 corresponds to 'no pain', score:10 corresponds to excessive pain)
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 2 weeks prior to intra-articular injection
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC), Score ranges between 0-100, Higher scores represent worse pain and poorer functioning, WOMAC score:0 corresponds to no functional impairment, WOMAC score:100 represents to complete impairment.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | at 2nd week following intra-articular injection
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC), Score ranges between 0-100, Higher scores represent worse pain and poorer functioning, WOMAC score:0 corresponds to no functional impairment, WOMAC score:100 represents to complete impairment.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | at 4th week following intra-articular injection
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC), Score ranges between 0-100, Higher scores represent worse pain and poorer functioning, WOMAC score:0 corresponds to no functional impairment, WOMAC score:100 represents to complete impairment.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | at 6th week following intra-articular injection
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC), Score ranges between 0-100, Higher scores represent worse pain and poorer functioning, WOMAC score:0 corresponds to no functional impairment, WOMAC score:100 represents to complete impairment.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Acıbadem Kozyatağı Hospital, Istanbul, Kozyatağı
  - Kartal Lutfi Kırdar State Hospital, Istanbul
  - Nevşehir State Hospital, Nevşehir

IPD SHARING:
Plan to Share IPD: Yes
Even recruitment has been closed this study is still on progress. We are willing the share all our available data for future studies.
Supporting Information: Study Protocol
Time Frame: Study Protocol will be available following the paper has been published.

REFERENCES:
- [Background] Jevsevar DS, Shores PB, Mullen K, Schulte DM, Brown GA, Cummins DS. Mixed Treatment Comparisons for Nonsurgical Treatment of Knee Osteoarthritis: A Network Meta-analysis. J Am Acad Orthop Surg. 2018 May 1;26(9):325-336. doi: 10.5435/JAAOS-D-17-00318. PMID 29688920
- [Background] Jayaram P, Kennedy DJ, Yeh P, Dragoo J. Chondrotoxic Effects of Local Anesthetics on Human Knee Articular Cartilage: A Systematic Review. PM R. 2019 Apr;11(4):379-400. doi: 10.1002/pmrj.12007. Epub 2019 Mar 15. PMID 30676699
- [Background] Busse P, Vater C, Stiehler M, Nowotny J, Kasten P, Bretschneider H, Goodman SB, Gelinsky M, Zwingenberger S. Cytotoxicity of drugs injected into joints in orthopaedics. Bone Joint Res. 2019 Mar 2;8(2):41-48. doi: 10.1302/2046-3758.82.BJR-2018-0099.R1. eCollection 2019 Feb. PMID 30915209
- [Background] Bellamy JL, Goff BJ, Sayeed SA. Economic Impact of Ketorolac vs Corticosteroid Intra-Articular Knee Injections for Osteoarthritis: A Randomized, Double-Blind, Prospective Study. J Arthroplasty. 2016 Sep;31(9 Suppl):293-7. doi: 10.1016/j.arth.2016.05.015. Epub 2016 May 18. PMID 27402605

DOCUMENTS (1):
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05291793/ICF_000.pdf